CLINICAL TRIAL: NCT02148445
Title: Smoking Cessation Versus Long-term Nicotine Replacement Among High-risk Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Edward Ellerbeck, MD, MPH, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000666; CER-1306-02901 (Other: PCORI)
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Smoking; Pulmonary Disease, Chronic Obstructive; Tobacco Use Disorder
Keywords: smoking cessation; tobacco use cessation products; nicotine
MeSH Terms: conditions — Smoking; Pulmonary Disease, Chronic Obstructive; Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Smoking Cessation (Active Comparator): Participants in the standard smoking cessation (SC) arm will receive a standard approach to smoking cessation, including smoking cessation counseling supplemented with 10 weeks of combination nicotine replacement therapy (NRT) (nicotine patch plus choice of gum or lozenge) if they are willing to make a quit attempt.
  Interventions: Other: Standard Smoking Cessation; Drug: Nicotine replacement therapy
- Extended Nicotine Replacement Therapy (Experimental): Participants in the guided maintenance therapy (GMT) arm will receive counseling focused on medication adherence and smoking reduction plus up to 52 weeks of combination nicotine replacement therapy (NRT) (nicotine patch plus choice of gum or lozenge) regardless of their interest in quitting.
  Interventions: Other: Extended Nicotine Replacement Therapy; Drug: Nicotine replacement therapy

INTERVENTIONS:
Other: Standard Smoking Cessation — Participants in the standard smoking cessation (SC) arm will receive a standard approach to smoking cessation, including smoking cessation counseling supplemented with 10 weeks of combination nicotine replacement therapy (NRT) (nicotine patch plus choice of gum or lozenge) if they are willing to make a quit attempt.
  Arms: Standard Smoking Cessation
Other: Extended Nicotine Replacement Therapy — Participants in the guided maintenance therapy (GMT) arm will receive counseling focused on medication adherence and smoking reduction plus up to 52 weeks of combination nicotine replacement therapy (NRT) (nicotine patch plus choice of gum or lozenge) regardless of their interest in quitting.
  Arms: Extended Nicotine Replacement Therapy
Drug: Nicotine replacement therapy
  Other Names: nicotine patch, nicotine gum, nicotine lozenge

SUMMARY:
Long-term NRT has not been studied in patients with COPD, and smokers in the United States with COPD are still asked to choose between immediate quitting or continued smoking. The purpose of this study is to see if guided maintenance therapy (GMT), using long-term NRT, might prove to be a reasonable alternative to the standard approach of asking patients to quit immediately. The investigators believe that GMT with long-term NRT will reduce overall exposure to cigarette smoke, reduce harm related to smoking, and ultimately lead to greater quit rates.

In this study, 398 smokers with COPD will be randomly assigned to either receive: 1) traditional smoking cessation (SC) or 2) long-term, guided maintenance therapy with NRT (GMT). The SC intervention will be based on a standard approach to smoking cessation, including smoking cessation counseling supplemented with combination NRT (a nicotine patch plus the patient's choice of gum or lozenge) if they are willing to make a quit attempt. The GMT intervention will consist of counseling, focused on medication adherence and smoking reduction, plus 52 weeks of combination NRT. After 3, 6 and 12 months of treatment, we will compare the two treatments based on their effects on smoking cessation, number of cigarettes smoked, exposure to carbon monoxide and smoking-related carcinogens, COPD symptoms, breathing function, and smoking-related hospitalizations or death. The investigators will also analyze the data in such a way that will be able to identify which patients are most likely to benefit from treatment. This analysis will allow patients to estimate their chances of success based on their own personal characteristics and which treatment they choose.

The investigators study addresses research priorities identified in recent smoking cessation guidelines and builds upon the input of our Patient Advisory Panel and our Stakeholder Advisory Committee. This study reflects the interests expressed by smokers in prior surveys and addresses the limited reach and effectiveness of traditional approaches to smoking cessation. If our GMT approach is effective, our study could change the recommendations provided in clinical practice guidelines and change the way that insurance companies pay for smoking cessation treatment. GMT could provide an alternative for millions of smokers with COPD who are not currently benefiting from traditional approaches to smoking cessation

DETAILED DESCRIPTION:
BACKGROUND Smokers with chronic obstructive pulmonary disease (COPD) recognize the dangers of continued smoking and would like to quit, but for most of them the idea of going 'cold turkey' is too intimidating. Many of these smokers would like to cut back on the amount that they smoke as part of a longer term path to quitting. Long-term nicotine replacement therapy (NRT) might allow them to do this. Long-term NRT is safe; it can reduce the rewarding effects of cigarettes, reduce the amount that people smoke, and increase quit rates. Long-term NRT has not, however, been studied in patients with COPD, and smokers in the United States with COPD are still asked to choose between immediate quitting or continued smoking. The purpose of this study is to evaluate the relative benefits of a third option: guided maintenance therapy with long-term NRT. We believe that long-term NRT could reduce overall exposure to cigarette smoke, reduce harm related to smoking, and ultimately lead to greater quit rates.

OBJECTIVES

1. Compare the benefits of traditional smoking cessation (SC) versus guided maintenance therapy (GMT) with NRT for smokers with COPD.
2. Estimate rates of smoking cessation and other patient-desired outcomes based on patient-specific characteristics and treatment choice (SC or GMT).

METHODS In this study, we will randomize 398 smokers with COPD to one of two treatment arms: 1) traditional smoking cessation (SC) or 2) long-term, guided maintenance therapy with NRT (GMT). Participants in the SC arm will receive a standard approach to smoking cessation, including smoking cessation counseling supplemented with combination NRT (nicotine patch plus choice of gum or lozenge) if they are willing to make a quit attempt. Participants in the GMT arm will receive counseling focused on medication adherence and smoking reduction plus 52 weeks of combined NRT. Outcomes will be measured at 3, 6 and 12 months post-randomization and will assess rates of smoking cessation, number of cigarettes smoked, exposure to carbon monoxide and smoking-related carcinogens, and clinical outcomes including respiratory symptoms, respiratory function, and smoking-related hospitalizations or death. In addition to directly comparing outcomes in the two treatment arms, our novel classification and regression tree analysis will allow us to identify subgroups of patients most likely to benefit from treatment and will allow patients to estimate their projected outcomes given their personal history and their choice of therapy.

PATIENT OUTCOMES (PROJECTED) This study will show how long-term NRT compares to a traditional smoking cessation program in helping smokers quit, reduce cigarette exposure, lower exposure to carcinogens, and reduce risk for death and hospitalizations. If our hypothesis is correct, this program could dramatically alter treatment choices for the millions of smokers in the United States with COPD that have been frustrated in their attempts to quit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Physician-diagnosed COPD
* Smoke 5 or more cigarettes/day
* Smoke cigarettes on 25 or more of the last 30 days
* Speak either English or Spanish
* Willing to take nicotine replacement therapy for up to 1 year and participate in study procedures

Exclusion Criteria:

* Reside in a facility that does not allow smoking
* Don't have an address and telephone
* Unstable cardiac condition (e.g. unstable angina or myocardial infarction in the past 30 days)
* Pregnant or breastfeeding
* Terminal illness with less than 12 month life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Ellerbeck, MD, Principal Investigator — University of Kansas
Locations (1):
- Kansas University Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will create a clean, de-identified copy of our dataset. It will be available to other researchers, upon request. We will make data available to users under a data sharing agreement that provides for (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Data will be saved as SAS or SPSS files, saved to disk, encrypted, and mailed to users. A copy of our analytic code used to generate our primary outcomes paper(s) will also be available on request. Given that this study does not meet the threshold for data sharing requirements, the costs of data preparation and shipping will be borne by the requester.

REFERENCES:
- [Derived] Ellerbeck EF, Nollen N, Hutcheson TD, Phadnis M, Fitzgerald SA, Vacek J, Sharpe MR, Salzman GA, Richter KP. Effect of Long-term Nicotine Replacement Therapy vs Standard Smoking Cessation for Smokers With Chronic Lung Disease: A Randomized Clinical Trial. JAMA Netw Open. 2018 Sep 7;1(5):e181843. doi: 10.1001/jamanetworkopen.2018.1843. PMID 30646142

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 667 Screened for Eligibility 153 Did not meet inclusion criteria 116 Refused to participate 398 Randomized
Period: Overall Study
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Started | 198 | 200
Completed | 197 | 197
Not Completed | 1 | 3
Not completed — Death | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy | Total
Number analyzed (Participants) | 198 | 200 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (8.66) | 55.7 (9.88) | 55.9 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 127 | 238
  Male | 87 | 73 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 190 | 195 | 385
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 35 | 82
  White | 113 | 123 | 236
  More than one race | 35 | 42 | 77
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 198 | 200 | 398
Number of Quit Attempts in the Past 12 Months [Mean (Standard Deviation); unit: number of quit attempts] | 2.2 (5.09) | 1.9 (4.29) | 2.1 (4.70)
Cigarettes Smoked per Day [Mean (Standard Deviation); unit: cigarettes per day] | 22.1 (11.87) | 24.0 (12.58) | 23.0 (12.26)
Carbon Monoxide Exposure [Mean (Standard Deviation); unit: parts per million] | 22.2 (13.12) | 22.7 (14.48) | 22.5 (13.81)
Carcinogen Exposure (Creatinine Adjusted NNAL) [Mean (Standard Deviation); unit: pg/mg] | 451.3 (422.74) | 507.4 (764.95) | 475.0 (604.41)
Number of respiratory-related hospital admissions and ED visits in the past 12 months [Count of Participants; unit: Participants]
  0 Visits | 122 | 134 | 256
  1 Visit | 30 | 36 | 66
  2 or more Visits | 46 | 30 | 76
Number of cardiac-related hospital admissions and ED visits in the past 12 months [Count of Participants; unit: Participants]
  0 Visits | 178 | 171 | 349
  1 Visit | 7 | 17 | 24
  2 or more Visits | 13 | 12 | 25
Respiratory Symptoms [Mean (Standard Deviation); unit: units on a scale] — Respiratory Symptoms as measured by the COPD Assessment (CAT) Test. This questionnaire measures the impact of Chronic Obstructive Pulmonary Disease (COPD) on well-being and daily life. Scores range from 0-40, with higher scores indicating higher levels of impact.
  units on a scale | 21.1 (8.82) | 22.9 (8.32) | 22.0 (9.00)
Respiratory Function [Mean (Standard Deviation); unit: % of predicted] — As measured by spirometry, FEV1
  % of predicted | 57.3 (18.61) | 56.7 (21.03) | 57.0 (19.84)
Cotinine [Mean (Standard Deviation); unit: ng/mg of creatinine] | 2395.8 (2184.80) | 2447.2 (2433.58) | 2421.6 (2310.39)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence (Point Prevalent)
Description: 7-day point prevalent abstinence at 12 months, confirmed by exhaled CO <=10
Time Frame: Month 12
Population: n=4 deceased participants were excluded from analysis. Missing values were counted as smokers.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
Participants | 23 | 24
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority — Based on prior studies using precessation NRT, we estimate a 2-fold increase in cessation outcomes in the GMT group compared to the SC group. Given our recruitment of patients at all levels of readiness to quit, we estimate a 12 month cessation rate of 10%. With 199 participants, in each arm, we will have an 80% power to detect a 2-fold difference or greater with a Type I error rate of 5%; p = 0.88, Chi-squared

2. Secondary Outcome: Sustained Abstinence
Description: 6 month sustained abstinence as measured by self-report at 6 and 12 months and confirmed by CO at 6 and 12 months. Participants who were confirmed as non-smokers by carbon monoxide (CO) at both Month 6 and Month 12 were considered to have "6-month sustained abstinence."
Time Frame: Month 6 through Month 12
Population: n=4 deceased participants were excluded from analysis. Missing values were counted as smokers.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
Participants | 15 | 12
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority — Based on prior studies using precessation NRT, we estimate a 2-fold increase in cessation outcomes in the GMT group compared to the SC group. Given our recruitment of patients at all levels of readiness to quit, we estimate a 12 month cessation rate of 10%. With 199 participants, in each arm, we will have an 80% power to detect a 2-fold difference or greater with a Type I error rate of 5%. This sample size will provide comparable power for looking at 6 month sustained cessation; p = 0.55, Chi-squared

3. Secondary Outcome: Quit Attempts
Description: Number of self-reported quit attempts over one year. At Month 3 and Month 6, participants reported the number of quit attempts in the last 3 months. At Month 12, participants reported the number of quit attempts in the last 6 months.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants were excluded from analysis.
Measure: Mean (Standard Deviation); unit: number of quit attempts
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
number of quit attempts
  Month 3: number analyzed (Participants) | 189 | 191
  Month 3 | 4.6 (6.54) | 3.7 (5.48)
  Month 6: number analyzed (Participants) | 181 | 185
  Month 6 | 4.5 (6.86) | 4.8 (8.97)
  Month 12: number analyzed (Participants) | 185 | 183
  Month 12 | 5.7 (8.59) | 6.2 (11.31)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.40, Mixed Models Analysis

4. Secondary Outcome: Average Cigarettes Per Day
Description: Average number of cigarettes per day over one year. Participants were asked at Month 3, Month 6, and Month 12 "During the past 7 days, on those days that you smoked, what was the average number of cigarettes or little cigars smoked per day?"
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants excluded from analysis
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
cigarettes per day
  Month 3: number analyzed (Participants) | 189 | 191
  Month 3 | 7.9 (8.64) | 10.5 (8.64)
  Month 6: number analyzed (Participants) | 182 | 185
  Month 6 | 8.1 (8.52) | 9.1 (9.45)
  Month 12: number analyzed (Participants) | 186 | 185
  Month 12 | 8.5 (7.84) | 8.1 (8.33)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.05, Mixed Models Analysis

5. Secondary Outcome: Carbon Monoxide Exposure
Description: Carbon monoxide (CO) exposure over 12 months. At Month 3, Month 6, and Month 12, participants completed an expired carbon monoxide laboratory test, which measured CO in parts per million.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants excluded from analysis
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
parts per million (ppm)
  Month 3: number analyzed (Participants) | 174 | 185
  Month 3 | 15.0 (12.62) | 17.4 (13.69)
  Month 6: number analyzed (Participants) | 164 | 167
  Month 6 | 14.6 (11.85) | 15.4 (12.58)
  Month 12: number analyzed (Participants) | 175 | 176
  Month 12 | 15.5 (11.14) | 13.8 (11.14)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.05, Mixed Models Analysis

6. Secondary Outcome: Carcinogen Exposure
Description: Creatinine-adjusted NNAL (4-(methylnitrosamino)-1-(3)pyridyl-1-butanol)) exposure over 12 months. At Month 3, Month 6, and Month 12, participants provided a urine sample that was used to assess their level of urinary creatinine and NNAL.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants were excluded from analysis.
Measure: Geometric Mean (Standard Deviation); unit: pg/mg creatinine
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
pg/mg creatinine
  Month 3: number analyzed (Participants) | 188 | 190
  Month 3 | 279.0 (353.42) | 320.1 (350.59)
  Month 6: number analyzed (Participants) | 180 | 184
  Month 6 | 178.2 (221.26) | 186.0 (236.21)
  Month 12: number analyzed (Participants) | 183 | 180
  Month 12 | 190.4 (233.22) | 183.5 (223.94)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.39, Mixed Models Analysis

7. Secondary Outcome: Respiratory Function
Description: Change in respiratory function, as measured by spirometry (FEV1), at 12 months post-randomization.
Time Frame: Month 12
Population: n=4 deceased participants excluded from analysis. Participants with missing data excluded.
Measure: Mean (Standard Deviation); unit: % of predicted
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 175 | 175
% of predicted | 55.4 (19.25) | 56.8 (19.78)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.42, t-test, 1 sided

8. Secondary Outcome: Respiratory Symptoms
Description: Respiratory symptoms as measured by the COPD Assessment Test (CAT) respiratory questionnaire. Participants completed this 8-item assessment at Month 3, Month 6, and Month 12. Scores range from 0 to 40, with higher levels indicating higher impact of COPD on well-being and daily life.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants excluded from analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
units on a scale
  Month 3: number analyzed (Participants) | 189 | 191
  Month 3 | 17.8 (9.25) | 19.3 (8.68)
  Month 6: number analyzed (Participants) | 181 | 185
  Month 6 | 17.9 (9.48) | 18.1 (8.51)
  Month 12: number analyzed (Participants) | 185 | 184
  Month 12 | 17.5 (9.33) | 18.2 (9.37)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.27, Mixed Models Analysis

9. Secondary Outcome: Respiratory-related Hospital Visits
Description: Number of respiratory-related hospital admissions and emergency room visits. Participants were asked how many times they had visited the ED or were admitted to the hospital for respiratory-related problems at Month 3, Month 6, and Month 12
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants excluded from analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
Participants
  Month 3: number analyzed (Participants) | 189 | 191
  Month 3: 0 Visits | 176 | 169
  Month 3: 1 Visit | 11 | 15
  Month 3: 2 or more Visits | 2 | 7
  Month 6: number analyzed (Participants) | 181 | 185
  Month 6: 0 Visits | 152 | 154
  Month 6: 1 Visit | 22 | 24
  Month 6: 2 or more Visits | 7 | 7
  Month 12: number analyzed (Participants) | 185 | 183
  Month 12: 0 Visits | 157 | 153
  Month 12: 1 Visit | 18 | 20
  Month 12: 2 or more Visits | 10 | 10
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.06, Mixed Models Analysis

10. Secondary Outcome: Cardiac-related Hospital Visits
Description: Number of cardiac-related hospital admissions and emergency room visits. Participants were asked how many times they had visited the ED or were admitted to the hospital for cardiac-related problems at Month 3, Month 6, and Month 12.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants excluded from analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
Participants
  Month 3: number analyzed (Participants) | 189 | 191
  Month 3: 0 Visits | 181 | 185
  Month 3: 1 Visit | 7 | 6
  Month 3: 2 or more Visits | 1 | 0
  Month 6: number analyzed (Participants) | 181 | 185
  Month 6: 0 Visits | 171 | 180
  Month 6: 1 Visit | 10 | 4
  Month 6: 2 or more Visits | 0 | 1
  Month 12: number analyzed (Participants) | 185 | 182
  Month 12: 0 Visits | 175 | 167
  Month 12: 1 Visit | 8 | 12
  Month 12: 2 or more Visits | 2 | 3

11. Secondary Outcome: 7-day Abstinence
Description: Self-reported and biochemically verified 7-day abstinence. Participants were asked at Month 3, Month 6, and Month 12, "Have you smoked any cigarettes or little cigars, even a puff, in the past 7 days?" They also completed an exhaled carbon monoxide lab test at Month 3, 6 and 12. Biochemical verification= exhaled CO <=10 ppm. Month 12 biochemically verified abstinence is the primary outcome, and is not reported in this table.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants were excluded from analysis. Missing responses were coded as smokers.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
Participants
  Month 3, self-report | 27 | 16
  Month 3, biochemically verified | 25 | 14
  Month 6, self-report | 28 | 20
  Month 6, biochemically verified | 25 | 19
  Month 12, self-report | 25 | 28
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Month 3 self-reported abstinence; Test type: Superiority; p = 0.08, Chi-squared
Statistical Analysis 2: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Month 3 biochemically verified abstinence; Test type: Superiority; p = 0.06, Chi-squared
Statistical Analysis 3: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Month 6, self-reported abstinence; Test type: Superiority; p = 0.22, Chi-squared
Statistical Analysis 4: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Month 6, biochemically verified abstinence; Test type: Superiority; p = 0.34, Chi-squared
Statistical Analysis 5: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Month 12, self-reported abstinence; Test type: Superiority; p = 0.66, Chi-squared

12. Secondary Outcome: Cotinine
Description: Cotinine over 12 months, adjusted for creatinine. At Month 3, Month 6, and Month 12, participants provided a urine sample that was used to assess their level of urinary creatinine and cotinine.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants were excluded from analysis
Measure: Geometric Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
ng/mg creatinine
  Month 3: number analyzed (Participants) | 188 | 190
  Month 3 | 2652.5 (2675.18) | 3378.1 (3182.00)
  Month 6: number analyzed (Participants) | 180 | 184
  Month 6 | 2390.7 (2842.07) | 3342.3 (3282.48)
  Month 12: number analyzed (Participants) | 183 | 180
  Month 12 | 2159.0 (2989.46) | 2363.7 (2988.16)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.0149, Mixed Models Analysis

13. Secondary Outcome: Average Cigarettes Per Day (Continued Smokers Only)
Description: Average number of cigarettes per day over one year, among continued smokers. All participants were asked "During the past 7 days, on those days that you smoked, what was the average number of cigarettes smoked per day?" at Month 3, Month 6, and Month 12. This analysis looks at the number of cigarettes per day among participants who were still smoking.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants excluded from analysis, non-smokers at each time point excluded
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
cigarettes per day
  Month 3: number analyzed (Participants) | 166 | 167
  Month 3 | 8.7 (8.84) | 11.4 (8.53)
  Month 6: number analyzed (Participants) | 159 | 161
  Month 6 | 9.1 (8.62) | 9.9 (9.52)
  Month 12: number analyzed (Participants) | 163 | 161
  Month 12 | 9.7 (7.64) | 9.3 (8.27)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.05, Mixed Models Analysis

14. Secondary Outcome: Carbon Monoxide Exposure (Continued Smokers Only)
Description: Carbon monoxide (CO) exposure over 12 months. At Month 3, Month 6, and Month 12, participants completed an expired carbon monoxide laboratory test, which measured CO in parts per million. This analysis looks at CO among those continuing to smoke.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants excluded from analysis, non-smokers at each time point excluded
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
parts per million (ppm)
  Month 3: number analyzed (Participants) | 152 | 161
  Month 3 | 16.4 (12.56) | 18.8 (13.23)
  Month 6: number analyzed (Participants) | 142 | 143
  Month 6 | 16.0 (11.68) | 17.0 (12.49)
  Month 12: number analyzed (Participants) | 153 | 152
  Month 12 | 17.4 (10.57) | 15.8 (10.73)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.08, Mixed Models Analysis

15. Secondary Outcome: Carcinogen Exposure (Continued Smokers Only)
Description: Creatinine-adjusted NNAL (4-(methylnitrosamino)-1-(3)pyridyl-1-butanol)) exposure over 12 months. At Month 3, Month 6, and Month 12, participants provided a urine sample that was used to assess their level of urinary creatinine and NNAL. This analysis looks at NNAL among continuing smokers only.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants were excluded from analysis, non-smokers at each time point excluded
Measure: Geometric Mean (Standard Deviation); unit: pg/mg creatinine
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
pg/mg creatinine
  Month 3: number analyzed (Participants) | 165 | 166
  Month 3 | 314.6 (373.23) | 337.6 (363.80)
  Month 6: number analyzed (Participants) | 158 | 160
  Month 6 | 219.8 (236.30) | 217.1 (251.82)
  Month 12: number analyzed (Participants) | 160 | 156
  Month 12 | 257.0 (234.83) | 247.5 (230.64)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.77, Mixed Models Analysis

16. Secondary Outcome: Cotinine (Continued Smokers Only)
Description: Cotinine over 12 months, adjusted for creatinine. At Month 3, Month 6, and Month 12, participants provided a urine sample that was used to assess their level of urinary creatinine and cotinine. This analysis looks at NNAL among continuing smokers only.
Time Frame: Month 3, Month 6, Month 12
Population: n=4 deceased participants were excluded from analysis, non-smokers at each time point excluded
Measure: Geometric Mean (Standard Deviation); unit: ng/mg creatinine
Groups:
- Standard Smoking Cessation: Participants in the standard smoking cessation (SC) arm will receive a standard approach to smoking cessation, including smoking cessation counseling supplemented with 10 weeks of combination nicotine replacement therapy (NRT) (nicotine patch plus choice of gum or lozenge) if they are willing to make a quit attempt.
  Standard Smoking Cessation: Participants in the standard smoking cessation (SC) arm will receive a standard approach to smoking cessation, including smoking cessation counseling supplemented with 10 weeks of combination nicotine replacement therapy (NRT) (nicotine patch plus choice of gum or lozenge) if they are willing to make a quit attempt.
  Nicotine replacement therapy
- Extended Nicotine Replacement Therapy: Participants in the guided maintenance therapy (GMT) arm will receive counseling focused on medication adherence and smoking reduction plus up to 52 weeks of combination nicotine replacement therapy (NRT) (nicotine patch plus choice of gum or lozenge) regardless of their interest in quitting.
  Extended Nicotine Replacement Therapy: Participants in the guided maintenance therapy (GMT) arm will receive counseling focused on medication adherence and smoking reduction plus up to 52 weeks of combination nicotine replacement therapy (NRT) (nicotine patch plus choice of gum or lozenge) regardless of their interest in quitting.
  Nicotine replacement therapy
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
Number analyzed (Participants) | 197 | 197
ng/mg creatinine
  Month 3: number analyzed (Participants) | 165 | 166
  Month 3 | 2771.2 (2774.24) | 3305.8 (2859.90)
  Month 6: number analyzed (Participants) | 158 | 160
  Month 6 | 2850.7 (2645.50) | 3502.2 (2978.67)
  Month 12: number analyzed (Participants) | 160 | 156
  Month 12 | 2733.9 (2532.32) | 2782.7 (2583.60)
Statistical Analysis 1: Comparison: Standard Smoking Cessation vs Extended Nicotine Replacement Therapy; Test type: Superiority; p = 0.0918, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Standard Smoking Cessation | Extended Nicotine Replacement Therapy
All-Cause Mortality (participants affected / at risk) | 1/198 | 3/200
Serious Adverse Events (participants affected / at risk) | 9/198 | 8/200
Other Adverse Events (participants affected / at risk) | 97/198 | 163/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Smoking Cessation (N=198) | Extended Nicotine Replacement Therapy (N=200)
Arrhythmia (Cardiac disorders) | 1 (1) | 3 (3) — Arrhythmia resulting in hospitalization or placement/modification of a device, but not a pacemaker for bradycardia
Hospitalization for CHF (Cardiac disorders) | 2 (2) | 2 (2) — Hospitalization for Congestive Heart Failure
Mesenteric Ischemia (Cardiac disorders) | 0 (0) | 1 (1) — Mesenteric Ischemia with death
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) — Myocardial Infarction would require hospitalization with elevated troponin
TIA (Cardiac disorders) | 1 (1) | 1 (1) — TIA with hospitalization
Revascularization (Cardiac disorders) | 3 (3) | 0 (0) — Revascularization - either a CABG or angioplasty/stent due to increasing ischemia
Stroke (Cardiac disorders) | 1 (1) | 0 (0) — Stroke with signs of sustained neurologic dysfunction
Unstable angina (Cardiac disorders) | 1 (1) | 0 (0) — Unstable angina requiring hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Smoking Cessation (N=198) | Extended Nicotine Replacement Therapy (N=200)
Local skin reactions (Product Issues) | 44 (89) | 81 (184) — Local skin reactions from the nicotine patch
Upper GI symptoms (Product Issues) | 32 (42) | 62 (89) — Including heartburn, indigestion, nausea, upset stomatch
Sleep Disturbance (Product Issues) | 23 (25) | 41 (51) — Including problems sleeping or vivid dreams
Oral discomfort (Product Issues) | 13 (14) | 26 (31) — Including sore throat, pain, blisters in mouth or jaw, dry mouth
Headache (Product Issues) | 7 (10) | 18 (21)
Change in affect or state of arousal (Product Issues) | 12 (13) | 20 (31) — including feeling jittery, nervous, anxious, restless, irritable, experiencing depressed mood, tiredness, sleepiness, fatigue
Cardiovascular symptoms (Product Issues) | 7 (9) | 13 (17) — Including change in blood pressure, heart rate, not a major cardiac event (MACE)
Hiccups (Product Issues) | 7 (8) | 11 (15)
Muscle Aches (Product Issues) | 1 (1) | 6 (8)
Bad Taste in Mouth (Product Issues) | 4 (5) | 11 (13) — Often reported as "nicotine taste in mouth"
Dizziness (Product Issues) | 3 (3) | 11 (11)
Increased Sweating (Product Issues) | 0 (0) | 7 (8) — Including night sweats
Diarrhea (Product Issues) | 4 (5) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No